CLINICAL TRIAL: NCT06690034
Title: Relationship of Serum Zinc Level with Severity of Diabetic Nephropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma kamal Eldin Mohamed Sayed, resident doctor at nephrology unit ,internal medicine department, Assiut University
Other Study IDs: Zinc and diabetic nephropathy
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Nephropathy Type 2
Keywords: serum zinc level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1: Patient with Diabetic kidney disease according to KDIG
- group 2: patients with diabetes without chronic kidney disease

SUMMARY:
Zinc influences the production and action of erythropoietin (EPO), a hormone produced by the kidneys that stimulates red blood cell production.

However, further research is needed to fully understand the mechanisms and to develop evidence-based guidelines for zinc supplementation in patient with Diabetic kidney disease. this study aim to detect serum zinc level in patient with Diabetic kidney disease "CKD" and Study of association between serum zinc and serum urea, creatinine, GFR, hemoglobin ,HbA1c in DKD

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is an irreversible , progressive disease with high morbidity and mortality that occurs commonly in the general adult population, especially in people with diabetes and hypertension . It's defined as decreased kidney function shown by glomerular filtration rate (GFR) of less than 60 mL/min per 1·73 m2, or markers of kidney damage, or both, of at least 3 months duration, regardless of the underlying cause .

Diabetic kidney disease represents the most common cause of CKD in developed countries. Approximately 30% to 40% of diabetes mellitus (DM) subjects develop Diabetic kidney disease "DKD", and its presence significantly increases the risk for morbidity and mortality.

Zinc is an essential element and is the second most abundant divalent cation in the human body (2-4 g). It is mainly distributed in skeletal muscles (57%) and bone (29%) and acts as a cofactor for more than 300 enzymes. In addition, zinc is involved in the cellular mechanisms of proliferation, maintenance of structural integrity, and in the systemic regulation of the immune system . Zinc seems to have a potential role in kidney and body homeostasis in diabetic individuals which include stabilization of insulin hexamers and pancreatic insulin storage and improved glycemic control. Decreased zinc levels can impair insulin function and glucose metabolism, potentially worsening diabetes control and increasing the risk of kidney damage. Zinc is important for maintaining endothelial cell integrity and function. Endothelial dysfunction is a hallmark of DKD, and decreased zinc levels can exacerbate vascular complications associated with diabetes. Lower serum zinc levels have been associated with increased proteinuria, a common symptom of DKD. Proteinuria indicates kidney damage and is a predictor of disease progression. Zinc is involved in modulating the immune response. Deficiency can lead to a heightened inflammatory state, exacerbating kidney damage. Several studies underline the critical role of zinc in reducing oxidative stress levels, which is considered the common denominator of the mechanisms responsible for the progression of kidney disease. Zinc is a cofactor for various enzymes involved in heme synthesis and erythropoiesis

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic kidney disease

Exclusion Criteria:

* patients on dialysis. Patient refuse to participate
* Other renal disease "lupus nephritis,GlomeruloNephritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic kidney disease and Diabetic patient without kidney disease as a control
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
zinc level | baseline
  prevalence of hypozincemia in Diabetic kidney disease

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Takao T, Yanagisawa H, Suka M, Yoshida Y, Onishi Y, Tahara T, Kikuchi T, Kushiyama A, Anai M, Takahashi K, Wakabayashi Sugawa S, Yamazaki H, Kawazu S, Iwamoto Y, Noda M, Kasuga M. Synergistic association of the copper/zinc ratio under inflammatory conditions with diabetic kidney disease in patients with type 2 diabetes: The Asahi Diabetes Complications Study. J Diabetes Investig. 2022 Feb;13(2):299-307. doi: 10.1111/jdi.13659. Epub 2021 Oct 7. PMID 34533892